CLINICAL TRIAL: NCT01506518
Title: Double Push Acoustic Radiation Force (DP ARF) Ultrasound for Monitoring Muscle Degeneration in Duchenne Muscular Dystrophy
Brief Title: Double Push Acoustic Radiation Force (DP ARF) Ultrasound for Monitoring Degeneration in Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11-1509; 1R01NS074057 (NIH)
Record Dates: First submitted 2011-12-22; First posted 2012-01-10 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-05

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Muscular Dystrophy, Duchenne; Ultrasound; Imaging; Acoustic Radiation Force; Double Push
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Duchenne muscular dystrophy and age 5-6 years: Boys diagnosed with Duchenne muscular dystrophy and age 5-6 years at enrollment.
- Duchenne muscular dystrophy and age 7-8 years: Boys diagnosed with Duchenne muscular dystrophy and age 7-8 years at enrollment.
- Duchenne muscular dystrophy and age 9-10 years: Boys diagnosed with Duchenne muscular dystrophy and age 9-10 years at enrollment.
- No known neuromuscular disorders and age 5-14 years: Volunteer boys ages 5-14 years with no known neuromuscular disorders to serve as controls.

SUMMARY:
This is a pilot clinical trial to assess the ability of a new ultrasound-based imaging method, Double-Push Acoustic Radiation Force (DP ARF) ultrasound, to monitor the progression of Duchenne muscular dystrophy. The hypothesis being tested is that DP ARF ultrasound delineates changes in muscle composition and function in individual dystrophic muscles, from early through late stages of disease development, that correlate to time to loss of ambulation in patient volunteers.

DETAILED DESCRIPTION:
Double Push Acoustic Radiation Force (DP ARF) imaging will be performed in 3 cohorts of up to 10 boys with DMD and in age-matched boys with no known neuromuscular disorders.

The first DMD cohort will enroll at age 5-6, the second at age 7-8, and the third at age 9-10. The rectus femoris (RF), cranial sartorius (CS), gastrocnemius (GAST), and lateral deltoid (DT) muscles will be targeted for their known phenotypic variation in response to dystrophin deficiency. The RF undergoes early necrosis and fatty deposition, the CS is thought to be relatively spared, and the GAST seems to undergo true hypertrophy. The DT, which undergoes hypertrophy like the GAST, will also be examined to determine if the impact of dystrophin deficiency varies between upper and lower limbs. All boys will be imaged 3 times annually for 4 years. In addition to DP ARF imaging every 4 mos, the boys will undergo standard quantitative muscle testing (QMT) and timed function tests (TFT) of time to standing, 6-minute walk, and 30-feet walk. Age at loss of ambulation will also be recorded for each boy. Boys with DMD generally loose ambulation by age 10, so we expect that the 20 boys in the 7-11 and 9-13 aged cohorts will lose ambulation over the course of this study. The 10 boys in the 5-9 aged cohort will likely not lose ambulation during the study. Because the primary objective of this clinical investigation is to evaluate the potential of DP ARF imaging as a relevant surrogate for monitoring disease progression and response to therapies, the focus of the study will be on correlating DP ARF results to change in functional degeneration and time to loss of ambulation.

There are two experimental components to this study beyond what is standard practice for DMD patients: 1) DP ARF ultrasound imaging of the rectus femoris (RF), cranial sartorius (CS), gastrocnemius (GAST), and lateral deltoid (DT) muscles and 2) standard quantitative muscle testing (QMT) and timed function tests (TFTs) of time to standing, 6-minute walk, and 30-feet walk repeated every four months (three times annually) throughout the four-year duration of the study.

This study will commence with DP ARF ultrasound imaging in the Clinical Neurophysiology Laboratory during the patient volunteer's first regularly scheduled research visit. Patient volunteers are expected to be outpatients. However, if a patient volunteer is an inpatient, DP ARF ultrasound imaging may be performed at the patient volunteer's hospital bedside. Immediately following DP ARF examination, the patient volunteer will undergo QMT and TFTs in the Physical Therapy Department. QMT and TFT will be conducted by trained physical therapists. DP ARF ultrasound imaging, QMT and TFT will be repeated as described above at each of the patient volunteers' twelve regularly scheduled research visits over the four-year study duration. Whenever possible, we will schedule research visits to coincide with other clinical visits to UNC. The patients' parents or caregivers will be compensated $50 per visit to defray the costs of travel to UNC, parking and lunch.

DP ARF will also be performed in 30 boys ages 5-14 with no known neuromuscular disorders. Imaging will be performed as described for the boys with DMD. The DP ARF results obtained in boys with no known neuromuscular disorders will be compared to those obtained in boys with neuromuscular disorders to serve as a control for changes in muscle mechanical property to occur with normal muscle growth and development.

DP ARF ultrasound is a noninvasive diagnostic imaging technology performed using commercially available clinical ultrasound imaging equipment - the Siemens Acuson Antares imaging system equipped for research purposes and VF10-5 or VF7-3 linear array transducers (Siemens Medical Solutions, USA Inc. Ultrasound Division). DP ARF imaging will be carried out by a professional sonographer, faculty and/or graduate student research assistants in the UNC-CH Joint Department of Biomedical Engineering. The sonographer will acquire DP ARF ultrasound data with matched B-Mode (for anatomical reference) in the right RF, CS, GAST, and DT muscles of patient volunteers. Patient volunteers will be asked to lie on an examination table in the Clinical Neurophysiology Clinic (outpatients) or to remain in their hospital beds (inpatients). The head of the exam table/bed may be raised to an approximate 45 degree angle to best visualize the muscles of interest with ultrasound imaging.

Once the patient volunteer is positioned, ultrasound gel will be applied to the patient volunteer's skin surface above the muscles of interest. The ultrasound imaging transducer will then be placed on top of the gel. Once the first muscle of interest is located, DP ARF ultrasound imaging will begin. We will orient the transducer to acquire ultrasound data transverse to the muscle fibers in the middle of the muscle length-wise, with three repeated acquisitions. We will then rotate our transducer 90 degrees to orient the imaging plane parallel to the muscle fibers. The previously imaged cross-section will be positioned in the approximate middle of the imaging field of view, with three repeated acquisitions. Muscle fiber orientation will be approximate, as surmised from anatomy. The DP ARF axial focal depth will be directed to the center of the muscle, approximately 20 - 30 mm.

The length of time for DP ARF data collection in each muscle is estimated to be less than 10 minutes. Once DP ARF imaging is completed on one muscle, DP ARF imaging will be performed on the other muscles of interest. Once all 4 muscles (RF, CS, GAST and DT) are imaged, the study procedure will be completed for the DP ARF imaging portion of the study.

For the second part of the study, beginning shortly (less than 4 hours) after DP ARF imaging is completed, the patient volunteer will undergo clinically standard quantitative muscle testing (QMT) of maximum voluntary isometric contraction (MVIC) in the right RF, CS, GAST and DT. The patient volunteer will also undergo clinically standard timed function tests (TFTs) of (1) time to rise from supine to standing, (2) distance walked in six minutes and (3) time to walk 30 feet.

Patient volunteers' participation will end once both study parts one (DP ARF ultrasound imaging) and two (QMT and TFT) are completed twelve times over 4 years. Therefore, there will be regularly scheduled follow-up visits required of the patient volunteers every four months. The patient volunteer is asked to assent and his parents are asked to permit their son to undergo (1) DP ARF ultrasound imaging of his right RF, CS, GAST and DT muscles, and (2) QMT and TFTs of time to standing, 6-minute walk, and 30-feet walk. No additional procedures or requirements are proposed. Every other aspect of the patient volunteers' care for DMD will be carried out in the normal standard of care as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Duchenne muscular dystrophy with clinical onset by age 5
* Ability to stand, alone or with assistance, at time of enrollment
* Ability to communicate with pertinent staff
* Ability to understand and comply with study requirements
* Ability to give informed consent.

Exclusion Criteria:

* Confirmed diagnosis of other muscle disease
* Previous compartment syndrome
* Previous injury to selected limbs
* Previous vascular surgery to selected limbs
* History of a compressive neuropathy (e.g., sciatic, femoral or tibial palsy in leg)
* History of rhabdomyolysis

Ages: 5 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include patient volunteers with Duchenne muscular dystrophy (DMD). Thirty volunteers (boys with DMD, enrolling at ages 5 (n=10), 7 (n=10), or 9 (n=10)) having clinical diagnosis of DMD with clinical onset by age 5 will be considered for enrollment.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change in DP ARF marginal peak displacement | once every 4 months for 4 years for 12 total measures
  Marginal peak displacement (MPD) is a metric developed to qualitatively describe the degree of nonlinearity in the viscoelastic properties of tissue: MPD = (P2-D)/P1, where P1 and P2 are the first and second peak displacement achieved in tissue by the first and second ARF excitations, respectively, and d is the ARF-induced displacement remaining at the time of the second push.

SECONDARY OUTCOMES:
Rate of change in DP ARF marginal peak displacement | 4 months to 4 years
  rates of change in marginal peak displacement will be measured from time-point to time-point (every 4 months) and across multiple time points (spanning 8 months to 4 years).
Change in quantitative muscle testing score of maximum voluntary isometric contraction (MVIC) | every 4 months for 4 years
  standard quantitative muscle testing of maximum voluntary isometric contraction (MVIC) in the rectus femoris, cranial sartorius, gastrocnemius, and lateral deltoid muscles of the right limbs.
Change in time to rise from supine position to standing | every 4 months for 4 years
  standard time to standing timed function test
Change in distance walked in six minutes | every 4 months for 4 years
  standard six-minute walk timed function test
Change in time to walk 30 feet | every 4 months for 4 years
  standard 30-feet walk timed function test
Rate of change in maximum voluntary isometric contraction (MVIC) | 4 months to 4 years
  rate of change in maximum voluntary isometric contraction (MVIC) will be assessed from time-point to time-point (4 month separation between measures) and across time-points (8 months to 4 years time separation between measures).
Rate of change in time to rise from supine to standing position | 4 months to 4 years
  rate of change in time to standing timed function test score will be assessed from time-point to time-point (4 month separation between measures) and across time-points (8 months to 4 years time separation between measures).
Rate of change in distance walked in six minutes | 4 months to 4 years
  rate of change in six-minute walk timed function test score will be assessed from time-point to time-point (4 month separation between measures) and across time-points (8 months to 4 years time separation between measures).
Rate of change in time to walk 30 feet | 4 months to 4 years
  rate of change in 30-feet walk timed function test score will be assessed from time-point to time-point (4 month separation between measures) and across time-points (8 months to 4 years time separation between measures).
Age at loss of ambulation | 4 years
  Loss of ambulation will be diagnosed by the patient volunteer's physician. The patient volunteer's age at the time loss of ambulation is first diagnosed will be recorded.
Change in percent degenerative muscle composition | every 4 months for 4 years
  Muscle boundaries will be hand-delineated using matched B-Mode image guidance in DP ARF marginal peak displacement parametric images. Within each 2D muscle image, percent degenerative area (Ad) will be calculated as T/N, where N is the total muscle area (number of pixels x area/pixel) and T is the muscle area in which marginal peak displacement values are within thresholds for necrosis, fat or fibrous tissue identification.
Change in percent necrotic tissue area | every 4 months for 4 years
  Muscle boundaries will be hand-delineated using matched B-Mode image guidance in DP ARF marginal peak displacement parametric images. Within each 2D muscle image, percent necrotic area (An) will be calculated as n/N, where N is the total muscle area (number of pixels x area/pixel) and n is the muscle area in which marginal peak displacement values are within thresholds for necrosis.
Change in percent fat tissue area | every 4 months for 4 years
  Muscle boundaries will be hand-delineated using matched B-Mode image guidance in DP ARF marginal peak displacement parametric images. Within each 2D muscle image, percent fatty deposition area (Af) will be calculated as f/N, where N is the total muscle area (number of pixels x area/pixel) and f is the muscle area in which marginal peak displacement values are within thresholds for fat tissue identification.
Change in percent fibrotic tissue area | every 4 months for 4 years
  Muscle boundaries will be hand-delineated using matched B-Mode image guidance in DP ARF marginal peak displacement parametric images. Within each 2D muscle image, percent degenerative area (Ac) will be calculated as c/N, where N is the total muscle area (number of pixels x area/pixel) and c is the muscle area in which marginal peak displacement values are within thresholds for fibrous tissue identification.

CONTACTS AND LOCATIONS:
Overall Officials: Caterina M Gallippi, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill Hospitals, Chapel Hill, North Carolina, United States